CLINICAL TRIAL: NCT02138305
Title: Collaborative Pilot Study to Determine the Correlation Between Intra-Operative Observations Using SPY® Near Infra-Red Imaging and Cardiac Catheterization Laboratory Physiological Assessment of Lesion Severity (PERSEUS Pilot Study)
Brief Title: Correlation Study of Imaging Data Acquired During CABG With Data Acquired in the Cath Lab
Acronym: PERSEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Volcano Corporation (Industry); Imperial College London (Other)
Responsible Party: Principal Investigator, Dr Ashesh N. Buch, Assistant Professor Cardiovascular Sciences (Interventional Cardiology), East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCIRB 13-001949; PERSEUS I (Other Grant/Funding Number: Volcano Corporation 120313)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve (FFR); Instantaneous Wave Free Ratio (iFR); Coronary Flow Reserve (CFR); Hyperemic Stenosis Resistance Index (HSR); Hyperemic microvascular resistance (HMR); Wave intensity analysis (WIA); Myocardial Perfusion; SPY NIRF Regional Myocardial Perfusion Analysis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Controlled prospective observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients referred for CABG (Other): * Patients who after undergoing standard of care diagnostic coronary angiography will be referred for CABG
  * ComboMap XT Guidewire
  * 'SPY' NIRF During CABG
  Interventions: Device: ComboMap XT Guidewire; Procedure: 'SPY' NIRF During CABG

INTERVENTIONS:
Device: ComboMap XT Guidewire — Intracoronary pressure and flow measurements
Procedure: 'SPY' NIRF During CABG — FDA approved use of injection of indocyanine green for the purposes of performing pre and post coronary grafting graft patency and perfusion assessment with the SPY near infra red fluorescence system

SUMMARY:
Visual assessment of a coronary artery narrowing (called stenosis) seen on angiography is conventionally used to infer how likely the stenosis will limit blood flow (called ischemia) under conditions of increased demand (e.g exercise). This is based on animal work and data from humans with simple single vessel disease with no co-existing conditions. These data have been extrapolated to more complex patients/ complex disease but clearly over-simplifies the situation in the majority of patients cardiologists treat.

Pivotal work by DeBruyne, Pils and colleagues in the 90's convincingly showed that pressure derived measurements, called FFR, from the coronary artery during a cardiac catheterization, more accurately identify stenoses that would cause ischemia compared to visual assessment alone. A strategy of FFR guided coronary stenting with drug eluting stents significantly improved outcomes and reduced costs compared to visual assessment alone (FAME trial). Deferring treatment based on FFR has been shown to be safe (DEFER Trial). FFR has excellent sensitivity and specificity. A FFR of <=0.80 was used as this identified ischemia causing lesions 90% of the time. Therefore, the concept of FFR guided percutaneous revascularisation and treatment deferral has a robust evidence base to support it.

Coronary bypass grafting (CABG) is traditionally based solely on a visual assessment of angiography images. SPY® Infrared Fluorescence Angiography (NIRF, FDA approved 2005) is used by some cardiac surgeons to assess the patency of bypass grafts in real-time in the operating room, as a surrogate for immediate traditional coronary angiography. Dr. Ferguson observed that regional myocardial perfusion (RMP) image data was also captured in these video sequences.

Study Hypotheses:

1. In patients who are likely CABG candidates, target vessel epicardial coronary arteries (TVECAs) with FFR > 0.80 will not demonstrate an increase in RMP despite an anatomically patent bypass conduit during SPY® imaging.
2. In TVECAs with an increase in RMP during SPY® imaging, cardiac catheter laboratory measures of coronary physiology from that TVECA, namely one or a combination of FFR, CFR, HSR and HMR, will correlate with the SPY® data on myocardial perfusion, and suggest a potential mechanism for this physiologic response to TVECA grafting.

ELIGIBILITY:
Inclusion Criteria:

* Age >18<80
* Patients with stable angina or NSTEMI with total CK rise of <1000 U/litre who after planned coronary angiography are going to be referred for CABG and have at least one vessel with a visual 40-80% stenosis that is interrogated with intracoronary physiology

Exclusion Criteria:

* Emergent status, or Cardiogenic shock
* LVEF <40%
* History of actively malignant disease
* Patient needing concomitant valvular surgery or other cardiac structural reconstructive surgery
* As is standard of care, those vessels that are extremely tortuous, very small caliber and/or heavily calcified would not have such wires passed down them. Furthermore, those vessels that are 80-90+% stenosed, with <TIMI 3 flow, which we would not normally pass a diagnostic physiology pressure wire, would not be studied with ComboXT wire.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12; Primary Completion 2018-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Correlation Analysis | 18 months
  Correlation between anatomy, functional anatomy, FFR, SPY® RMP change, and the presence or absence of imaged competitive flow

OTHER OUTCOMES:
Correlation Analysis | 18 months
  Correlation analysis between anatomy, functional anatomy, FFR, CFR, HMR and SPY® perfusion data for each TVECA and perfusion territory.
Instantaneous Wave Free Ratio (iFR) | 18 months
  Offline analysis of de-identified encrypted data for each TVECA interrogated with ComboMap XT wire by Dr Justin Davies's research group, Imperial College, London for iFR determination. Correlation analysis between iFR and presence or absence of imaged competitive flow and intra-operative RMP data on SPY® NIRF
Wave Intensity Analysis (WIA) | 18 months
  Offline wave wave intensity analysis (WIA) of de-identified encrypted data for each TVECA interrogated with ComboMap XT wire by Dr Justin Davies's research group, Imperial College, London. Correlation analysis between WIA data and presence or absence of imaged competitive flow and intra-operative RMP data on SPY® NIRF

CONTACTS AND LOCATIONS:
Overall Officials: Ashesh N Buch, MBChB, MD, Principal Investigator — East Carolina University; T. Bruce Ferguson, MD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina Heart Institute at Vidant Medical Center, Greenville, North Carolina, United States